CLINICAL TRIAL: NCT04126603
Title: Impact of Semaglutide (Long Acting GLP1 Agonist) on Peripheral Blood Derived CD34+ Endothelial Cells (EPCs) and Subcutaneous Fat Derived Mesenchymal Stromal Cells ( MSCs) in Type 2 Diabetes Subjects
Brief Title: Impact of Semaglutide on CD34+ EPC and Fat Derived MSC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sabyasachi Sen (Other)
Responsible Party: Sponsor-Investigator, Sabyasachi Sen, Professor of Medicine, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCR191206
Record Dates: First submitted 2019-10-07; First posted 2019-10-15 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A Placebo (Placebo Comparator): Placebo.
  Interventions: Drug: Placebos
- Group B Active (Active Comparator): Semaglutide
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — 0.25mg/week for week 0 - 4 , then increasing to 0.5mg/week for weeks 5 - 8, then 1 mg/week for week 9 - 24 weeks
  Arms: Group B Active
Drug: Placebos — Placebo injection
  Arms: Group A Placebo

SUMMARY:
The Investigator is trying to ascertain whether an FDA approved medication of T2DM, Semaglutide, can improve the number, function and gene expression of subjects CD34+ endothelial progenitor cells. EPCs are the source of cells protecting the inner lining of blood vessels and improving their survivability will improve cardiovascular outcome as high glucose environment of diabetes are toxic to these EPC Cells.

Improve mitochondrial metabolism of Mesenchymal Stem Cell from subcutaneous fatty tissue, leading to weight loss. Improve overall vascular health by reducing inflammation.

The investigator will enroll 40 subjects with T2DM who are only on metformin. The study consists of 4 visits to the GW MFA, including screening visit. Subjects will be recruited from across the DMV area, and prescreened over the phone or in clinic, and then invited for an in-person screening visit at the GW MFA to determine eligibility. If eligible, subject will be enrolled into one of two study Arms, active semaglutide 1 mg or Placebo. This study will include an up titration of study drug. From week 0-4 subject will be on 0.25 mg/week, from week 5-8 subject will take 0.5mg/week, and week 9 to 24 subject will take 1 mg/week of Semaglutide or Placebo.

During the regular 3 visits subject will have their vital measured, body composition assessed using Tanita scale, arterial stiffness measured and blood drawn for EPC cells analysis and standard of care labs. At visit 1 and visit 3, fat biopsy will be done on the belly area to acquire 2-3 grams of fat tissue. Screening will take place at week -2, Visit1 at week 0, Visit 2 at week 8, Visit 3 at week 24. Subject will receive follow-up phone calls on week 4, week16 and week 28.

DETAILED DESCRIPTION:
Diabetes affects more than 9% of adults in the United States and this is projected to nearly double by 2025. Both diabetes and obesity are associated with endothelial dysfunction, oxidative stress, endothelial cell inflammation, cardiovascular pro-thrombotic states and are the most common causes of kidney disease and blindness. Endothelium and its progenitors, meaning endothelial progenitor cells (EPCs), are an established surrogate of cardiovascular risk outcome measures. EPCs have been defined as CD34+ cells thereby identifying a defined homogenous population from a heterogeneous peripheral blood derived mononuclear cells.

The investigator and others, have previously shown that EPCs can act as a cellular biomarker that is more reliable than serum based markers for CVD risk estimation. It was demonstrated that gene expression in EPCs change within two weeks of an intervention such as aerobic exercise. On the other-hand serum biomarkers usually take much longer time to change secondary to an intervention. Also the paracrine effect of damaged endothelium is secondary to gene expression changes that have been altered in the progenitor cells several months ahead of discernible changes in serum based biomarkers such as endothelium based inflammatory markers. When serum inflammatory markers are elevated that may mean that the endothelium is already damaged/ inflamed and possibly irreversibly

EPC are the future endothelium, therefore studying EPCs may help us to predict the effect of an intervention (such as a medication or exercise) on the future of endothelium and endothelial function. In normal course of events, the EPCs transition to mature endothelium and replace endothelial cells after normal cell death cycle or programmed apoptosis. However, unfortunately, type 2 diabetes being a pro-inflammatory, high ROS disease process, chronically depletes the EPC population by up-regulating apoptotic pathways mediated by p53. As an apoptotic condition, hyperglycemia even mild (such as prediabetes) affects immature EPCs more so than the mature endothelium. Hence, the damaged and inflamed mature endothelium, with time, is not replaced by EPCs as the progenitor pool has been depleted. This maybe one of the reasons why vascular damage takes 4-5 years to develop following onset of hyperglycemia.

It is known that GLP1 agonist has positive effect on oxidative stress, and endothelial function, therefore semaglutide can be hypothesized to have a positive effect on EPC and endothelium and possibly reduce fat inflammation. It may also reduce transformation of multipotent mesenchymal stem cells (MSCs) towards more fat formation (prevent adipogenesis) which may explain weight reducing capability seen in semaglutide studies (SUSTAIN trials). The use of CD34+ cells and MSCs as a biomarker is novel. One can obtain CD34+ cells from a simple peripheral blood draw (without doing an invasive procedure). The blood is then sorted for a homogenous progenitor/stem cell population. Role of CD34+ve EPCs in vascular biology, heart regeneration and collateral vessel formation as an endothelial progenitor cell is well established. It's role as a biomarker is also being developed. CD34+ cells are the most studied cardiovascular progenitor cells and its efficacy has been established in chronic diseases such as diabetes by Werner et al in 2005.

Similarly, one can obtain fat derived MSC from fat biopsies, particularly from overweight and obese individuals. Diabetes is not only a state of endothelial dysfunction, it is also a state of fat hyperplasia, insulin resistance at the level of muscle and fat and is associated with high ROS. Improvement of endothelial health is most likely paired with healthier fat. A state of healthier fat will be associated with healthy adipocytes, pre-adipocytes and healthy MSCs.

The weight reducing data from SUSTAIN 6 trial using semaglutide at 0.5mg and 1.0mg, is encouraging. It has also shown significant improvement in blood pressure and HbA1C within 8 weeks and definitely by 16 weeks even at a lower FDA approved dose of 0.5mg once a week.

These finding prompted the investigator team to use MSC as a fat surrogate and EPCs as an endothelial surrogate to establish a cellular mechanism behind the clinical trial findings. It may also shed light on cross-talk between these two important insulin responsive tissues that contribute towards cardiovascular health.

The Investigators believe EPC is the ideal cellular vascular outcome biomarker while MSC is the ideal adipocyte health bio-marker. Based on recently published data on saxagliptin's effect on EPC of subjects with Type 2 Diabetes, the investigators are confident that EPC is a robust endothelial marker with quick changes in number, function and gene expression, after appropriate intervention.

The purpose of the present study is to study the effect of a long-acting GLP-1 agonist, over a period of 24 weeks and understand how it influences two different yet related cell types such as endothelium and adipocyte, both of which are key players in insulin resistance/sensitivity in the body.

Study Hypotheses:

The investigator hypothesize that GLP1 agonists, like semaglutide, have a positive effect on the EPC number, function, targeted gene expression, arterial stiffness and endothelium specific inflammatory markers.

Additionally, the investigator hypothesize that semaglutide therapy will reduce adipogenesis and increase bone and cartilage formation by increasing cellular metabolism, as evidenced by increased mitochondrial biogenesis and increased cellular oxygen consumption rate (OCR, measured by SeaHorse).

ELIGIBILITY:
Inclusion Criteria

* Age 20-90
* Diagnosed with Type 2 diabetes mellitus
* Body Mass Index (BMI) between 25.0-45.0 (both inclusive)
* eGFR ≥ 30 mL/min/1.73 m2 by MDRD
* HbA1C 6.5 - 12.0 %
* Subjects on lifestyle modification alone, or Metformin (0.5-2 grams), insulin, or in combination, in any doses of either Metformin or Insulin for at least 3 months prior to screening. 2 week washout of any other anti-hyperglycemic.
* Ability to provide informed consent (and document informed consent by signature) before any trial-related activities are conducted.
* Additional CVD risk factor such microalbuminuria or proteinuria (as defined by ADA, UACR > 30 mg/g), hypertension (labile, uncontrolled hypertension or controlled on anti-hypertensives) and left ventricular hypertrophy, left ventricular systolic or diastolic dysfunction, or an ankle brachial index [the ratio of the systolic blood pressure at the ankle to the systolic blood pressure in the arm] of less than 0.9, low HDL with hypertriglyceridemia (as defined by NCEP ATP III) , strong family history of CHD (as defined by NCEP ATP III and ATP IV).
* Retinal examination within last 2 years of enrollment, showing no proliferative retinopathy

Exclusion Criteria

* Uncontrolled hyperglycemia with fasting glucose >300 mg/dL (>16.6 mmol/L)
* Liver disease with ALT, AST or ALP ≥ x3 ULN
* Known (recent) personal history of cerebral stroke or heart attack (myocardial infarction) within last 6 months
* Personal or family history of medullary thyroid cancer (MTC)
* Personal or family history of Multiple Endocrine Neoplasia Syndrome Type 2 (MEN 2)
* GFR <30 mL/min/1.73 m2 by MDRD
* Prior surgery with chronic malabsorption (eg, bariatric) within last 1 year
* Clinically significant RBC disorders such as hemoglobinopathies
* Diagnosis of Type 1 diabetes mellitus or history of GAD antibody positive status
* Chronic use of high dose anti-inflammatory drugs for the last 3 months
* Beginning statin medications or change in statin dose within the past 1 month
* Starting use of high-dose steroid medication (100mg hydrocortisone or 40mg prednisone equivalent) within the last 1 month
* History of acute pancreatitis within the past 2 years
* Known or suspected allergy to GLP-1 agonists, excipients, or related products.
* Active smokers, >5 per day (at present)
* Any other clinical condition that would jeopardize patients safety while participating in this clinical trial
* Women of child bearing potential who are not willing to use a contraceptive method to avoid pregnancy for the 16 weeks of study duration plus 2 months post treatment (for semaglutide washout).
* Women who are pregnant or breastfeeding
* Chronic or persistent alcohol or drug abuse
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg. infectious disease) illness
* Participation in another trial with an investigational drug within 30 days prior to informed consent.
* Untreated or active hemorrhagic proliferative diabetic retinopathy

Exclusionary Laboratory Findings

* Chronic Kidney Disease (CKD) stage 5 (estimated CrCl less than 15 mL/min)
* Triglycerides > 500 mg/dL
* Low hematocrit (<28 Units)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2025-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Washington VA Medical Center, Washington D.C., District of Columbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients were enrolled at GWU
Pre-assignment Details: Only 10 patients from GWU were enrolled in the study.
Period: Overall Study
Arm/Group | Group A Placebo | Group B Active
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A Placebo: Metformin + Placebo.
  Placebos: Placebo injection
- Group B Active: Metformin + Semaglutide: 0.25mg/week for week 0 - 4 , then increasing to 0.5mg/week for weeks 5 - 8, then 1 mg/week for week 9 - 24 weeks
- Total: Total of all reporting groups
Arm/Group | Group A Placebo | Group B Active | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 59 [29 to 72] | 59 [53 to 73] | 59 [29 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 3 | 1 | 4
  More than one race | NA — not reported | NA — not reported | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: CD34+ Endothelial Progenitor Cell Number (EPC) Per Mononuclear Cells (MNC) Ratio
Description: Number of CD34+ EPCs per total MNC ratio. Please note CD34+ cells is a progenitor cell marker derived from mononuclear cells (MNCs).
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
ratio
  First visit | 0.10 (0.06) | 0.23 (0.16)
  Last visit | 0.12 (0.03) | 0.13 (0.09)

2. Primary Outcome: CD34+ Endothelial Progenitor Cell Migration (EPC) Against Serum SDF1a Gradient
Description: The distance the CD34+ EPC migrates in response to SDF1 alpha 10ng. This assess the mobility of stem cells such as CD34+ EPC and the distance it traveled would lead us to understand how medication therapy changes stem cell behavior and its functionality.
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: micrometer (um)
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
micrometer (um)
  First visit | 708.5 (357.09) | 377.75 (440.17)
  Last visit | 530.75 (405.53) | 3232.33 (2553.21)

3. Primary Outcome: Gene Expression of CD34+ Endothelial Progenitor Cell Number
Description: we will evaluate mRNA gene expression of endothelial Progenitor cell with catalase, KDR, NOS3,SOD2, TNF-alpha which is normalized to 18s. Fold change of particular genes in hematopoietic stem cells between baseline and terminal visit at week 24 were analyzed.
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
Fold change
  Catalase | -0.64 (0.72) | 0.5 (1.52)
  KDR | 0.78 (0.05) | 1.49 (0.43)
  NOS3 | -1.88 (0.05) | 2.33 (0.05)
  SOD2 | 0.56 (0.48) | 0.97 (0.69)
  TNF-A | 3.37 (2.75) | -1.09 (0.83)

4. Primary Outcome: CD34+ Endothelial Cell Colony Formation Unit (CFU)
Description: CFU count of CD34+ EPCs
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: CFUs/mL
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
CFUs/mL
  First Visit | 12.0 (4.77) | 5.10 (1.56)
  Last Visit | 12.25 (11.67) | 23.75 (4.60)

5. Secondary Outcome: Gene Expression of Subcutaneous Adipose Cell
Description: We will evaluate mRNA gene expression for mature fat and fat related transcription factors.
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Population: Due to freezer power failure in the lab, the fat samples were degraded and could not saved for cryo preservation. As a result, qpcr and histology could not carried out due to lack of samples in frozen state.
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Arterial Stiffness: Pulse Wave Analysis Augmentation Index
Description: Vessel health is assessed by looking at Arterial stiffness. Augmentation index (AI) is defined as the ratio of the augmentation pressure to the pulse pressure, times 100, to give a percentage. We used Vascular Flow and wave measurement equipment, SphygmoCor Central Pressure system from AtCor. The higher the values the higher the cardiovascular risk.
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
percent
  First visit | 23.80 (11.82) | 29.67 (4.16)
  Last visit | 24.00 (0.05) | 32.00 (14.14)

7. Secondary Outcome: Arterial Stiffness: Pulse Wave Analysis Augmentation Pressure
Description: Arterial Stiffness: Pulse Wave Analysis Augmentation Pressure. The higher the values the higher the cardiovascular risk.
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
Millimeters of mercury
  First visit | 10.80 (7.69) | 15.33 (2.89)
  Last visit | 8.00 (0.05) | 16.50 (13.44)

8. Secondary Outcome: Arterial Stiffness: Pulse Wave Analysis Augmentation Index 75
Description: Vessel health is assessed by looking at Arterial stiffness. Augmentation index (AI) is defined as the ratio of the augmentation pressure to the pulse pressure, times 100, to give a percentage. Augmentation index 75 normalizes this value to an estimate of the AI at a heart rate of 75bpm. We used Vascular Flow and wave measurement equipment, SphygmoCor Central Pressure system from AtCor. The higher the values the higher the cardiovascular risk.
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
percent
  First visit | 23.20 (15.80) | 32.00 (7.55)
  Last visit | 27.00 (0.05) | 36.50 (14.85)

9. Secondary Outcome: Body Composition: BMI
Description: Body mass index measured using Bio metric Impedance Scale
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: Kilogram per meter squared
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
Kilogram per meter squared
  First visit | 34.95 (4.68) | 44.33 (7.75)
  Last visit | 36.00 (6.32) | 40.77 (4.00)

10. Secondary Outcome: Body Composition: Body Fat Percent
Description: Percent of Body Fat measured using Bio metric Impedance Tanita Scale
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
percent
  First visit | 41.10 (5.98) | 50.70 (0.5)
  Last visit | 39.47 (9.09) | 49.87 (6.77)

11. Secondary Outcome: Biochemistry: Hemoglobin A1C (HbA1c)
Description: HbA1c percent
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
percent
  First visit | 7.67 (2.05) | 7.80 (1.27)
  Last visit | 6.55 (1.48) | 7.10 (0.57)

12. Secondary Outcome: Hip to Waist Ratio
Description: Ratio of Hip to Waist
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
Ratio
  First visit | 0.96 (0.2) | 0.94 (0.06)
  Last visit | 0.79 (0.1) | 0.95 (0.03)

13. Secondary Outcome: Biochemistry: Low-density Lipoprotein (LPL) Cholesterol Over High-density Lipoprotein (HDL) Ratio
Description: ratio of LDL over HDL cholesterol
Time Frame: First Visit at Baseline and Last Visit at 24 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Group A Placebo | Group B Active
Number analyzed (Participants) | 5 | 5
Ratio
  First visit | 2.43 (0.49) | 1.23 (0.55)
  Last visit | 1.98 (0.28) | 1.97 (0.74)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Patients monitored by laboratory results every 2 months and questions of general well-being
Arm/Group | Group A Placebo | Group B Active
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04126603/Prot_SAP_002.pdf
  • Informed Consent Form (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04126603/ICF_003.pdf